CLINICAL TRIAL: NCT02466659
Title: A Clinical Trial of Observation Versus Controlled Intermittent Alternate Occlusion (CIAO) Therapy for Intermittent Exotropia
Brief Title: Controlled Intermittent Alternate Occlusion (CIAO) Therapy for Intermittent Exotropia
Acronym: CIAO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no fund
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Principal Investigator, Daniel E. Neely, Professor of Ophthalmology, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IndianU
Record Dates: First submitted 2015-04-14; First posted 2015-06-09 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Intermittent Exotropia
Keywords: IXT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CIAO Therapy (Experimental): Intervention with wearing 3-hour daily CIAO therapy glasses
  Interventions: Device: CIAO therapy Amblyz glasses
- Observation (No Intervention): To observe as one kind of standard care for IXT.

INTERVENTIONS:
Device: CIAO therapy Amblyz glasses — 3-hour CIAO Therapy Amblyz glasses
  Arms: CIAO Therapy

SUMMARY:
To determine the effectiveness of alternate occlusion therapy for the treatment of IXT among patients aged 3 to < 11 years old.

DETAILED DESCRIPTION:
Intermittent exotropia (IXT) is the most common form of childhood-onset exotropia with an incidence of 32.1 per 100,000 in children. Before surgery, many cases of IXT are treated using non-surgical interventions, such as part-time alternate occlusion. However, the "alternating" occlusion with traditional patches is usually out of control. The investigators are uncertain about the amount of "alternating" in patching treatment.

Here, the investigators introduce controlled intermittent alternating occlusion (CIAO) therapy, which is provided by a new electronic device, -liquid crystal glasses. This study is to determine the effectiveness of alternate occlusion therapy for the treatment of IXT among patients aged 3 to < 11 years old. Children with IXT will be randomized into either an observation group or a CIAO therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent exotropia (manifest deviation) meeting all of the following criteria:

  * Intermittent exotropia at distance OR constant exotropia at distance and either intermittent exotropia or exophoria at near
  * Exodeviation at least 15PD at distance OR near measured by prism and alternate cover test (PACT)
  * Exodeviation at least 10PD at distance measured by PACT
* No previous surgical or non-surgical treatment for IXT (other than refractive correction)
* Visual acuity in the worse eye 0.3 logMAR or better (20/40 on ATS HOTV or 70 letters on E-ETDRS) for children ≥ 3 years of age
* No interocular difference of visual acuity more than 0.2 logMAR (2 lines on ATS HOTV or 10 letters on E-ETDRS) for children ≥ 7 years of age
* Investigator not planning to initiate amblyopia treatment
* No hyperopia greater than +3.50 D spherical equivalent in either eye
* No myopia greater than -6.00 D spherical equivalent in either eye
* No prior strabismus, intraocular, or refractive surgery
* No abnormality of the cornea, lens, or central retina
* Investigator willing to observe the IXT untreated for 3 years unless specific criteria for deterioration are met.

Exclusion Criteria:

* N/A

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Neely, MD, Principal Investigator — Glick Eye Institute
Locations (1):
- Glick Eye Institute, Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CIAO Therapy | Observation
Started | 5 | 3
Completed | 0 | 1
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CIAO Therapy | Observation | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: Year] | 5.7 (1.94) | 6.24 (4.17) | 5.91 (2.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
IXT Control Score at distance [Mean (Standard Deviation); unit: units on a scale] — IXT control score: referring to the Pediatric eye disease investigator group (PEDIG).
  PEDIG scale of control for IXT 1-5 is defined as the following:
  * 5 = Constant exotropia
  * 4 = exotropia > 50% of the 30-sec period before dissociation
  * 3 = exotropia < 50% of the 30-sec period before dissociation
  * 2 = No exotropia unless dissociated, recovers in > 5 sec
  * 1 = No exotropia unless dissociated, recovers in 1-5 sec
  * 0 = No exotropia unless dissociated, recovers in < 1 sec (phoria)
  * Not Applicable = No exotropia present
  units on a scale | 4 (.71) | 2.67 (.57) | 3.5 (.92)

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Measure of IXT Control Score
Description: IXT control score: referring to the Pediatric eye disease investigator group (PEDIG).
  PEDIG scale of control for IXT 1-5 is defined as the following:
  5 = Constant exotropia 4 = exotropia > 50% of the 30-sec period before dissociation 3 = exotropia < 50% of the 30-sec period before dissociation 2 = No exotropia unless dissociated, recovers in > 5 sec
  1 = No exotropia unless dissociated, recovers in 1-5 sec 0 = No exotropia unless dissociated, recovers in < 1 sec (phoria) Not Applicable = No exotropia present
Time Frame: 12 weeks; 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CIAO Therapy | Observation
Number analyzed (Participants) | 0 | 1
units on a scale |  | 5

2. Other Pre Specified Outcome: Amblyopia
Description: It is defined when visual acuity between two eyes equal or over 2 logMAR lines.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | CIAO Therapy | Observation
Number analyzed (Participants) | 0 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3MO
Arm/Group | CIAO Therapy | Observation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes